CLINICAL TRIAL: NCT05407350
Title: Validation of an Intestinal Ultrasound Score Evaluating Inflammation and Treatment Response in Crohn's Disease (USE-IT): A Prospective Multicenter Study
Brief Title: Validation of an IUS Activity Index
Acronym: USE-IT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: International Bowel Ultrasound Group e.V. (Other)
Responsible Party: Sponsor
Other Study IDs: USE-IT-01434
Record Dates: First submitted 2022-04-25; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-04

CONDITIONS: Crohn Disease
Keywords: intestinal ultrasound; MRE; Colonoscopy
MeSH Terms: conditions — Crohn Disease | interventions — Ultrasonography; Colonoscopy; Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Stuhl, Biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Crohns disease patients: Adult patients with moderately to severely active CD
  Interventions: Diagnostic Test: Ultrasound, Colonoscopy, MRE

INTERVENTIONS:
Diagnostic Test: Ultrasound, Colonoscopy, MRE — After the initiation of an established treatment of known efficacy for CD (biologic agents including infliximab, adalimumab, ustekinumab or vedolizumab either with or without corticosteroids), repeat IC and MRE will occur at Week 30 (± 6 weeks) (6-9 months); the IUS, IC, and MRE examinations will occur within a 4-week window and with no intervening change in medical therapy. All imaging data will be captured electronically (IUS and MRE with Digital Imaging and Communications in Medicine [DICOM] images, and IC with video recordings) for central, blinded reading. Two biopsies will be collected from each segment of the bowel (rectum, sigmoid, descending, transverse, ascending and terminal ileum) during IC, fixed in formalin collection containers, and shipped for histopathology processing and evaluation.
  Other Names: Collection of blood; Collection of Stuhl; Biopsie

SUMMARY:
The primary objective of this study is to prospectively validate a novel intestinal ultrasound (IUS) Crohn's disease (CD) activity index and component items, correlating CD activity and responsiveness to therapy as evaluated by IUS with evaluations by ileocolonoscopy (IC) (Simple Endoscopic Score for Crohn's disease [SES-CD]) and magnetic resonance enterography (MRE) (Simplified Magnetic Resonance Index of Activity [MaRIA] score).

DETAILED DESCRIPTION:
Study Design Prospective multicenter study of 111 participants with CD with 50 weeks of follow-up Study Population Adult patients with moderately to severely active CD

Inclusion Criteria:

1. Confirmed diagnosis of CD according to standard clinical, endoscopic, and histologic criteria of at least 3 months duration
2. Adults 18 years of age or older
3. Moderate to severely active CD defined by:

   1. Active symptoms with a HBI ≥ 8, and
   2. Bowel wall inflammation defined as bowel wall thickness (BWT) > 3 mm in at least 1 segment of the ileum or colon as determined by IUS
4. Patients with planned introduction of biologic therapy as per their treating gastroenterologist to treat active disease
5. Written informed consent must be obtained and documented

Exclusion Criteria:

1. Patients with a primary diagnosis of ulcerative colitis or IBD type unclassified
2. Patients with prior intestinal surgery
3. Patients with disease-related structural bowel complications, defined as either:

   1. Stricture with increased bowel wall thickening (>25% of normal), decreased luminal diameter (≥ 50% relative to the normal adjacent bowel loop) and proximal dilation (on any imaging modality), or
   2. Penetrating complications (excluding perianal fistulizing disease; patients with perianal disease are eligible if there is additional inflammation in another bowel segment [other than the rectum])
4. Contraindication to IC or MRE
5. BMI greater than 35 at time of screening or other characteristics considered likely to preclude IUS visualization of all bowel segments
6. Disease limited to the rectum
7. Serious underlying disease other than CD that in the opinion of the investigator may interfere with the participant's ability to participate fully in the study
8. History of alcohol or drug abuse that in the opinion of the investigator may interfere with the participant's ability to comply with the study procedures
9. Pregnancy Data Sources and Data Collection Data will be collected from patient charts (paper or electronic) including medical and CD related history, medication records, and results of prior laboratory and imaging examinations. Patient disease-related outcomes including hospitalizations, emergency department (ED) visits, and surgeries will be collected during visits for analysis. Data will be transcribed from the patient's chart and entered into an electronic case report form by the investigator or authorized trained designee.

Questionnaires are to be completed by healthcare professionals and patients (i.e., baseline demographics, HRQoL ]SIBDQ], PRO-2, IBD Knowledge Questionnaire).

Outcomes

Primary Outcome:

• The longitudinal and construct validity and treatment responsiveness of an IUS CD activity index in an adult population with moderate to severely active CD

Secondary Outcomes:

* The correlation of IUS CD activity index and component items with IC
* The correlation of IUS CD activity index and component items with MRE
* The correlation of IUS CD activity index and component items with biomarkers
* The correlation of IUS CD activity index and component items with clinical activity scores
* The correlation of IUS CD activity index and component items with histology
* The correlation of IUS CD activity index and component items with HRQoL (SIBDQ) and PRO-2
* The proportion of patients with IUS response and transmural healing after initiation of a biologic therapy approved for CD
* The longitudinal validity of changes in IUS CD activity and component items after treatment with changes in IC, MRE, biomarkers, clinical disease activity scores, HRQoL (SIBDQ), PRO-2, and histology
* The correlation of terminal ileal small bowel peristalsis with IUS CD activity index and component items, MRE, and IC with CD activity
* The correlation of IUS CD activity index and component items with patient outcomes, including ED visitation, hospitalization, and surgery.

Statistical Methods Demographic and clinical data will be evaluated using descriptive statistics. A putative IUS CD activity index in development using at least moderately reliable (inter-rater ICC > 0.40) items from a prior study (Part I) and its component items will be evaluated in this prospective cohort study.

Sample Size:

Power calculations are based on the primary endpoint of IUS CD activity index responsiveness. Based on the variance formula for the standardized mean change, and assuming a correlation of 0.3 for baseline and follow-up scores, a sample size of 94 paired scores would have 80% power to detect a standardized mean change of 0.35. Accounting for 15% attrition, a sample size of 111 participants will be needed.

Outcome Analysis:

The primary aim of this study is to both establish IUS CD activity index responsiveness to effective medical therapy with demonstration of changes in activity over time as well as index external validation through correlation of individual IUS activity index components and overall score compared to both IC and MRE.

Similar correlations will be examined between the IUS CD activity index and HBI, GHAS, RHI, SIBDQ, PRO-2, transmural healing, terminal ileal small bowel peristalsis, and patient outcomes including ED visitation, hospitalization, and surgery. All participants in this prospective cohort will receive medical therapy of known efficacy for CD. The definition of change will be based on a global IUS measure of disease activity, quantified using a 100 mm visual analog scale (VAS), where 0 represents no disease activity and 100 represents the worst disease activity ever seen. Clinically meaningful change will be defined by a decrease of more than ½ the SD of the global IUS VAS at Baseline. Longitudinal validity will be correlated with changes in the IUS CD activity index and other measures of disease activity on IC, and changes in MRE (Simplified MaRIA score), HBI, CRP, and fCal. Responsiveness will be quantified using the standardized effect size (mean difference divided by SD) and the associated 95% CI, as well as the nonparametric probability for detecting change, expressed as the AUROC. Weighted correlation coefficients will be used to quantify longitudinal validity. An exploratory knowledge questionnaire (IBD Knowledge Questionnaire) will also be used to evaluate the evolution of patient IBD understanding through study participation. The potential for this study data to be applied in machine learning IUS diagnostics will also be considered.

Expected Impact Development of a reliable and responsive IUS CD activity index will improve standardization and consistency in IUS utilization globally. In the long-term, this can profoundly change the way in which IBD care is delivered, with wider adoption of repeatable accurate disease activity evaluation in clinic resulting in accelerated uptake of a treat-to-target strategy in CD. This strategy has been demonstrated to better inform clinical decision making, improve patient outcomes, and reduce long-term disability in patients with CD. In addition, an increased IUS uptake can engage patients to better understand their disease which will result in improved adherence to monitoring and treatment which will ultimately improve CD related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CD according to standard clinical, endoscopic, and histologic criteria of at least 3 months duration
2. Adults 18 years of age or older
3. Moderate to severely active CD defined by:

   1. Active symptoms with a HBI ≥ 8, and
   2. Bowel wall inflammation defined as BWT > 3 mm in at least 1 segment of the ileum or colon as determined by IUS
4. Patients with planned introduction of biologic therapy as per their treating gastroenterologist to treat active disease
5. Written informed consent must be obtained and documented.

Exclusion Criteria:

1. Patients with a primary diagnosis of ulcerative colitis or IBD type unclassified
2. Patients with prior intestinal surgery
3. Patients with disease-related structural bowel complications defined as either:

   1. Stricture with increased bowel wall thickening (>25% of normal), decreased luminal diameter (>50% relative to the normal adjacent bowel loop) and proximal dilation (on any imaging modality) or;
   2. Penetrating complications (excluding perianal fistulizing disease; patients with perianal disease are eligible if there is additional inflammation in another bowel segment [other than the rectum]).
4. Contraindication to IC or MRE
5. BMI greater than 35 at time of screening or other characteristics considered likely to preclude IUS visualization of all bowel segments
6. Disease limited to the rectum
7. Serious underlying disease other than CD that in the opinion of the investigator may interfere with the participant's ability to participate fully in the study
8. History of alcohol or drug abuse that in the opinion of the investigator may interfere with the participant's ability to comply with the study procedures
9. Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a multicenter, international, nonrandomized prospective cohort study across multiple sites in North America, Australia, and Europe.
  The study population will consist of 111 adult participants with moderately to severely active CD managed as per SOC, in established IBD expert centers with access to IUS, IC, and MRE procedures.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The longitudinal and construct validity and treatment responsiveness of an IUS CD activity index in an adult population with moderate to severely active CD | week 0 to week 50
  The newly formed activity index determined by intestinal ultrasound is compared with the results of colonoscopy (IC), MRE, blood and stool markers.

SECONDARY OUTCOMES:
The correlation of IUS CD activity index and component items with IC | week 0 to week 50
  Disease activity determined by intestinal ultrasound is compared with the results of colonoscopy (IC) examinations.
The correlation of IUS CD activity index and component items with MRE | week 0 to week 50
  Disease activity determined by intestinal ultrasound is compared with the results of MRE examinations.
The correlation of IUS CD activity index and component items with biomarkers | week 0 to week 50
  Disease activity determined by intestinal ultrasound is compared with the results of Biomarker analysis.
The correlation of IUS CD activity index and component items with histology | week 0 to week 50
The correlation of IUS CD activity index and component items with HRQoL (SIBDQ) and PRO-2 | week 0 to week 50
  Disease activity determined by intestinal ultrasound is compared with the results of patient-reported outcomes HRQoL (SIBDQ) and PRO-2.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Novak, Prof, Principal Investigator — University of Calgary
Locations (1):
- IBUS office, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided